CLINICAL TRIAL: NCT00230581
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Multiple Doses and Dose Levels of DDP225 in Female Patients With Irritable Bowel Syndrome With Diarrhea
Brief Title: 8 Weeks Treatment With DDP225 in Patients With Diarrhea Predominant IBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dynogen Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDP225-04-006
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS-d, IBS
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

INTERVENTIONS:
Drug: DDP225

SUMMARY:
In this study, female patients with IBS-d will be treated for 8 weeks to assess the safety and effectiveness of DDP225 on GI transit and in reducing IBS symptoms.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multicenter study designed to assess the safety and efficacy of DDP225 in patients with IBS-d. Female patients from 18 to 65 years of age with a history of IBS-d for at least 6 months are potentially eligible for entry into the study. A total of 88 eligible patients with IBS-d will be studied.

The total duration of study participation for an individual patient is approximately 10 weeks (74 days) from the initial screening visit to final study evaluations. The total duration of dosing with study medication (either DDP225 or placebo) is 8 weeks.

Patients who satisfy all of the inclusion criteria and none of the exclusion criteria are eligible to enter the Treatment Period and will be randomly assigned to one of four treatment groups.

After a patient is randomized and enters the Treatment Period, she will take the appropriate study medication once a day for 56 days and return to the clinic at two week intervals for a total of four visits during the Treatment Period. During the Treatment Period, patients will maintain a daily diary and complete questionnaires. One week after completing the 56-day Treatment Period, patients return to the clinic for final safety evaluations which include a physical examination, electrocardiogram, and clinical laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients from 18 to 65 years of age, inclusive.
2. History of IBS-d for at least 6 months prior to the initial screening visit.
3. Endoscopic/radiologic bowel evaluation to rule out cancer, obstruction, or other structural disease.
4. The patient must have completed at least six days of assessments in the patient diary in the one week period prior to the second screening visit.
5. Negative serum and urine pregnancy tests and post-partum for at least one year or not breast feeding at the initial screening visit and throughout the study. For patients able to bear children, an acceptable method of birth control must be used throughout the study. Patients unable to bear children must have documentation of such in the case report form (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
6. Able to provide voluntary, written informed consent with comprehension of all aspects of the protocol.

Exclusion Criteria:

1. Serious underlying diseases, including psychiatric disorders or current history of conditions affecting bowel transit including biochemical or structural abnormalities, or GI surgery
2. Clinically significant abnormal examination findings or laboratory tests
3. Inability to stop taking certain medications, or a planned change in medication (including herbal remedies) which could interfere with study assessments
4. Use of drugs and or ethanol which may interfere with compliance of study procedures or influence study outcome
5. Presence of a medical condition which could interfere with the interpretation of study data
6. Significant use of nicotine or caffeine

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2005-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
GI Transit

SECONDARY OUTCOMES:
Patient Reported Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: William Patterson, MD, Study Chair — Hotel Dieu Hospital
Locations (16):
- United States (5):
  - Radiant Research, Scottsdale, Arizona
  - Radiant Research, St Louis, Missouri
  - Long Island Gastrointestinal Research, Great Neck, New York
  - Radiant Research, Mogadore, Ohio
  - Radiant Research, Greer, South Carolina
- Canada (11):
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - St. Joseph's Healthcare, London, Ontario
  - Meadowlands Family Health Centre, Ottawa, Ontario
  - London Road Diagnostic Clinic, Sarnia, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Toronto, Ontario
  - Hopital St-Sacrement, Québec, Quebec